CLINICAL TRIAL: NCT00158938
Title: Clinical Study of the EASYTRAK 3 Spiral Fixation Coronary Venous Bipolar Pace/Sense Lead
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Clinicals0007
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-06-25 (Estimated); Status verified 2007-06

CONDITIONS: Congestive Heart Failure
Keywords: Artificial Cardiac Pacemaker; Implanted Electrodes
MeSH Terms: conditions — Heart Failure

INTERVENTIONS:
Device: EASYTRAK 3 left ventricular pacing lead

SUMMARY:
The purpose of this clinical investigation was to assess the safety and effectiveness of the EASYTRAK 3 lead

DETAILED DESCRIPTION:
This clinical study was a prospective, multi-center, clinical evaluation to document safety and effectiveness of the EASYTRAK 3 lead in humans. Patients implanted with the EASYTRAK 3 lead were followed through pre-discharge, 1-month, 3-month and 6-month follow-ups

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe heart failure (NYHA Class III/IV) including left ventricular dysfunction (EF <= 35%) and QRS duration >= 120 ms remaining symptomatic despite stable, optimal heart failure drug therapy.
* Creatinine < 2.5 mg/dL obtained no more than two weeks prior to enrollment.
* Age 18 or above, or of legal age to give informed consent specific to state and national law.
* Willing and capable of providing informed consent, undergoing a device implant, participating in all testing associated with this clinical investigation at an approved clinical investigational center and at the intervals defined by this protocol.

Exclusion Criteria:

* A known hypersensitivity to a 1.0 mg (0.5 mg per electrode) dose of dexamethasone acetate.
* Previous cardiac resynchronization therapy, a coronary venous pace/sense lead or attempted LV lead placement.
* Pre-existing cardioversion/defibrillation leads other than those specified in this investigational plan (unless the investigator intends to replace them with permitted cardioversion/defibrillation leads).
* Requiring dialysis.
* A myocardial infarct, unstable angina, percutaneous coronary intervention, or coronary artery bypass graft during the preceding 30 days prior to enrollment.
* Hypertrophic obstructive cardiomyopathy or infiltrative cardiomyopathy (e.g., amyloidosis, sarcoidosis).
* A documented life expectancy of less than 6 months or expected to undergo heart transplant within 6 months.
* Enrolled in any concurrent study, without prior Guidant written approval, that may confound the results of this study.
* Have a mechanical tricuspid heart valve.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115
Dates: Start 2003-05; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Pacing thresholds at 6 months
Pacing impedances at 6 months
R-wave amplitudes at 6 months
6-month complication free rate

SECONDARY OUTCOMES:
left ventricular bipolar pacing and sensing with RENEWAL 3 H173 safety